CLINICAL TRIAL: NCT01170585
Title: A Randomised Placebo Controlled Trial of Rosuvastatin in Systemic Lupus Erythematosus
Brief Title: A Trial of Rosuvastatin in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-006214-16
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Atherosclerosis; Systemic Lupus Erythematosus
MeSH Terms: conditions — Atherosclerosis; Lupus Erythematosus, Systemic | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): randomised to placebo.
  Interventions: Drug: Placebo
- Active (Active Comparator): randomised to rosuvastatin.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — All patients will be uptitrated from an initial start dose of 5mg to 20mg rosuvastatin. This will be given once a day for 2 years.
  Other Names: Crestor
  Arms: Active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a condition that affects the whole body. It can cause inflammation of the blood vessels resulting in an earlier thickening and hardening of the arteries resulting in strokes. It has been reported that SLE can worsen the function resulting in heart failure.

The aim of the study is to examine what effects Rosuvastatin, a cholesterol lowering drug, given to patients has on the degree of thickening of the arteries over the course of two years. We also want to see how it affects the function of the blood vessels and also of the heart.

Individuals who agree to participate will be randomly assigned into two groups. One group will be given the active drug whereas the other will have a placebo. Subjects in the study will all have a cardiac magnetic resonance (CMR) scan before treatment, at 1 year and then 2 years at the end of the treatment. Each scan will involve imaging the carotid arteries in the neck, the arteries in the arm and also the heart. Individuals will continue to have regular out-patient reviews by their own team of doctors, regular blood tests will be taken to monitor the disease and also to ensure the safety and well being of the individual.

At the end of the 2 year study we hope that we will be able to slow down the rate of arterial thickening and retard any plaque build up in the arteries. We also want to see what effect rosuvastatin has on heart function. Ultimately, we hope to prove that people with SLE should be treated with a cholesterol lowering drug as part of their routine treatment.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an auto-immune condition, multisystem, connective tissue disorder with a wide spectrum of disease (D'Cruz et al 2007), which includes cardiovascular manifestations. It is a condition which primarily affects females with a predominance of 10:1. The peak onset is between 18 and 40 years of age. The incidence is reported to be higher amongst Asian and African ethnic groups. In the UK, the incidence is 3.8 per 100 000 per year, with a prevalence of 26.2 per 100 000. The incidence among the white UK population is 3.0 per 100 000 per year, whereas it is 10.0 among Asians and 21.89 among the Afro-Caribbean population, the highest of any population studied so far (Danchenko 2006). No clear aetiology has been identified, and the genetics are complex.

The range of cardiovascular manifestations is varied; it includes accelerated atherosclerosis, vascular inflammation (El-Magadmi, 2002) and ventricular dysfunction (Pieretti J, 2007). The presence of carotid atherosclerosis is a strong predictor of future cardiovascular events (Belcaro G, 1996) and as such, identification of plaque within the carotid arteries has been studied using ultrasound. Studies have also been conducted to investigate endothelial dysfunction and the relationship with SLE.

* Case studies of patients with SLE have shown patients with SLE have increased carotid intima-media thickness (IMT) on ultrasound (US) studies (Svenungsson E, 2001).
* US studies in SLE have reported endothelial dysfunction as demonstrated bu US flow mediated dilatation (FMD) (Lima DS, 2002, Celermaier DS, 1994).
* Ultrasound studies in SLE have demonstrated a significant correlation between dysfunctional endothelium (reduced flow-mediated dilatation/brachial artery reactivity) and carotid IMT (Raza K, 2000).
* Myocardial dysfunction, in particular, an increased left ventricular ejection fraction and mass due to left ventricular hypertrophy has been identified in this population (Chow PC, 2007, Pieretti J, 2007).

The excess cardiovascular risk in patients with SLE has been attributed to corticosteroid usage in the treatment of the condition and as such was given as the explanation of the increased atherosclerosis (Petri M, 1992, 1996). Although, corticosteroid therapy can itself cause hypertension, diabetes and dyslipidaemia, the cumulative steroid dose is also a surrogate marker for disease severity. Studies have also shown that patients with the condition are more hypertensive and have an increased tendency to be smokers (Asanuma Y, 2003). However, a separate study showed that despite a higher incidence of hypertension, diabetes and an earlier menopause, the 10 year Framingham risk score was the same as matched healthy controls (Bruce IN, 2003). This would suggest that the risk factors present in SLE are not adequately explained by the conventional cardiovascular risk assessment model. In fact, SLE itself is a strong independent risk factor for atherosclerosis. Due to the inflammatory nature of SLE it is consistent with the recent paradigm shift towards the concept of atherosclerosis as a disease of vascular inflammation. Vascular inflammation leads to endothelial and vascular damage which can predispose to atherosclerosis (Ross R, 1999).

The association of dyslipidemia and SLE has been demonstrated (Svenungsson E, 2001). There is elevation of LDL-cholesterol, triglycerides and lipoprotein (a)(Asanuma Y, 2003) with a decrease in HDL-cholesterol (Borba EF, 1994). Together with the elevation of alpha-1 anti-trypsin and homocysteine levels lead to conditions with are conducive for the development of atherosclerosis.

The mainstay of treatment of atherosclerosis in SLE is predominantly directed at controlling inflammation with aggressive conventional cardiovascular disease risk factor management with corticosteroids, anti-inflammatories and disease modifying drugs (cyclosporin A and azathioprine). For lipid management, it has been suggested that even in the absence of atherosclerosis, the LDL-cholesterol level should be <2.6mmol/L. However, there has been limited clinical data to demonstrate the benefit of this approach (Wajed J,2004, Bruce IN, 2005).

There has been much published data on the effect of lipid lowering drugs or statins (HMG-Co A reductase inhibitors) and plaque regression (Corti,2001, 2005, Lima J, 2004). These trials demonstrated a significant reduction in the amount of plaque within the vessel wall as well as the reduction of LDL-cholesterol. A recently published randomised placebo-controlled trial (METEOR) (Crouse J, 2007)showed that rosuvastatin 40mg once daily over 2 years arrested carotid plaque progression which continued in the placebo group. This study was was highly significant (P<0.01). In this study, carotid plaque and carotid intima media thickness (CIMT) was assessed by B-mode ultrasound. Such studies prove that there is a benefit of using statins in those with low risk or who have established plaque disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with SLE-as diagnosed by ACR criteria
* Male or females who are 18-80years of age, inclusive at screening
* Female subjects who are post menopausal (i.e >6mnths without menstrual period), surgically sterile, or using effective contraceptive measures at visit 0 and the same contraception throughout the study and for 30days after discontinuing treatment
* No current or previous statin therapy
* No current indication for statin therapy (Coronary artery disease; hypercholesterolemia, renal dysfunction)
* Subjects who have given their signed consent to participate in the study

Exclusion Criteria:

* Patient < 18 or > 80 years
* Contraindications for MRI - patients with pacemakers' defibrillators or pacing wires in the heart, or other metal implants such as metal in the eye, brain or spine. Other metallic devices or implants will have to be declared by the participant and assessed to be safe prior to having an MRI current or previous statin
* Known atherosclerotic valvular disease
* Renal dysfunction
* Hyperlipidemia
* Active myositis
* All forms of liver disease
* Pregnancy
* Breastfeeding
* Patients being treated with Cyclosporin A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in bilateral carotid artery wall volume and distensibility | 3 CMR of 24 months (baseline; 12 and 24 mnths)
  A series of 20 contiguous 2 dimensional images, centred about the carotid bifurcation will be obtained. These images are then used to calculate the vessel area, but because they are contiguous a three dimensional structure can be formed and the vessel volume can be calculated. These values can be plotted against age and sex-matched graphs of normal ranges.
  The carotid artery distensibility will be calculated by obtaining a short cine film of the carotid artery as it pulsates. This can be contoured in the diastolic and systolic phases of the cardiac cycle.

SECONDARY OUTCOMES:
Endothelial function assessed by brachial artery reactivity. | 3 CMR, baseline; 12 and 24 mnths.
  Endothelial function is assessed by imaging the area of the brachial artery at baseline & post intervention.Endothelial dependent function will be assessed by inflating a blood pressure cuff around the forearm for 5 minutes to occlude arterial blood flow and create hyperaemia on release which induces brachial artery dilation by shear effects on endothelium.Glyceryl trinitrate spray will be given to the patient, and further images will be obtained.Both sets of images will be compared to the baseline and the percentage change in vessel size calculated providing a measure of endothelial function.
Correlation of vascular findings to ventricular volumes and function | baseline; 12 and 24 months
  The correlation of ventricular indices in SLE patients is determined through assessment of cardiac function. Patients will have left and right ventricular volumes measured, allowing calculation of the ejection fraction. These will be compared with age and sex matched normal subjects

CONTACTS AND LOCATIONS:
Overall Officials: Dudley J Pennell, MD, Principal Investigator — CMR Unit, Royal Brompton Hospital, London
Locations (2):
- United Kingdom (2):
  - Imperial College NHS Trust, London, London
  - North West London Hospitals NHS Trust, London, London